CLINICAL TRIAL: NCT06061848
Title: Intralymphatic Immunotherapy Enhanced by Vitamin-D, a Randomized Placebo-controlled Trial and Comparison With SLIT
Acronym: ILIT vs SLIT
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Lars Olaf Cardell (Other)
Responsible Party: Sponsor-Investigator, Lars Olaf Cardell, Professor, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Dnr KS: K2021-5840
Record Dates: First submitted 2023-09-11; First posted 2023-09-29 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Allergic Rhinitis Due to Grass Pollen
MeSH Terms: interventions — Vitamin D; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- SLIT (Active Comparator): Sublingual immunotherapy timothy pollen 75000 SQ-T 1 daily for 3 years
  Interventions: Drug: SLIT Grazax ALK Nordic 75 000 SQ-T
- ILIT + Vitamin D (Active Comparator): Intramuscular injection of kolecalciferol 100000 IU followed by intralymphatic immunotherapy with 3 monthly injections of grass pollen allergen 1000 SQ-U.
  Interventions: Drug: ILIT + Vitamin D
- ILIT + placebo (Active Comparator): Intramuscular injection of saline solution followed by intralymphatic immunotherapy with 3 monthly injections of grass pollen allergen 1000 SQ-U.
  Interventions: Drug: ILIT + placebo

INTERVENTIONS:
Drug: SLIT Grazax ALK Nordic 75 000 SQ-T — Daily sublingual grass allergen tablets
  Arms: SLIT
Drug: ILIT + Vitamin D — 1 mL of Vicotrat D3, Heyl Pharma, 100 000 IU/mL, as intramuscular injection. Followed by 0,1 mL of Alutard SQ timothy, ALK Nordic, 10 000 SQ-U/mL as three intralymphatic injections
  Other Names: Alutard SQ timothy and Vicotrat D3
  Arms: ILIT + Vitamin D
Drug: ILIT + placebo — 1 ml of Sodium chloride solution 9 mg/mL as intramuscular injection followed by 0,1 mL of Alutard SQ timothy, ALK Nordic, 10 000 SQ-U/mL as three intralymphatic injections
  Other Names: Alutard SQ timothy and Sodium chloride
  Arms: ILIT + placebo

SUMMARY:
A national, multicenter, randmised double blind study with parallell arms. 360 patients with grass induced allergic rhinitis will be open randomised 1:2 to 3 years Grazax sublingual immunotherapy or 3 intralymphatic injections with ALK Alutard Timothy. In a second step, the ILIT group will be double blind randomised 1:1 to an intramuscular injection of Vitamin D Vicotrat or placebo, 4 week before the start of the intralymphatic treatment. The primary outcome measure is daily combined symptoms and medication scores during grass pollen season.

ELIGIBILITY:
Inclusion Criteria:

* moderate to severe allergic rhinitis due to grass pollen, with Rhinitis Total Symptom Score >/= 8.
* informed consent

Exclusion Criteria:

* chronic rhinosinusitis with or without nose polyps
* Previous immunotherapy (SLIT or SCIT)
* BMI > 35
* house dust mite allergy with symptoms
* allergy towards furry animals if exposition cannot be avoided
* 25(OH)Vitamin D levels < 25 or > 75 nmol/L
* use of Vitamin D supplementation or excessive use of sun tanning booths
* mental incapacity to follow study protocol
* other significant disease
* allergy towards study medication
* uncontrolled asthma
* severe atopic dermatitis
* pregnancy or nursing
* autoimmune disease
* hyper IgE-syndrome
* cardiovascular disease
* lung disease
* liver or kidney disease
* hematologic disorder
* metabolic disease
* chronic infectious disese
* medications interacting with the immune system
* cancer
* previous cytostatic therapy
* medication with beta-blockers or ACE-inhibiters, if medication cannot be paused at the day for treatment
* drug or alcohol abuse
* intake of other study product within 1 month or 6 half times, which ever is longest, before visit 1
* withdrawn consent

Exclusion Criteria only for ILIT group (due to vitamin D treatment)

* medication witch can interacts with vitD: (ACE-inhibitors, antiepileptic drugs, glycosides, orlistat, statines, thiazide diuretics)
* tendency for formation of kidney stones
* hyperparathyroidism or other disease conferring risk of hypercalcemia
* hereditary pseudohypoparathyroidism with decreased phosphorous secretion
* malabsorption or bowel disease with diarrhea
* Mb Paget, osteoporosis or sarcoidosis
* skin disease at the groin (where the treatment will be injected)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 360 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2030-12-28 (Estimated); Study Completion 2031-12-28 (Estimated)

PRIMARY OUTCOMES:
CSMS | 60-75 days at the grass pollen season year 1; 4 months before treatment. 60-75 days year 2; 6 months after start of treatment.
  Daily Combined Symptoms and Medication Scores (0-3)

SECONDARY OUTCOMES:
CSMS peak pollen season | 15 days at the grass pollen season year 1; 4 months before treatment. 15 days year 2; 6 months after start of treatment.
  Daily Combined Symptoms and Medication Scores (0-3) during the 15 consecutive days with the highest pollen count
RQLQ | 60-75 days at the grass pollen season year 1; 4 months before treatment. 60-75 days year 2; 6 months after start of treatment.
  Juniper Rhinoconjunctivitis Quality of Life Questionnaire, weekly scores (0-28)
VAS (0-10) | 4-6 months before treatment and 6-9 months after treatment
  Recalled symptoms severity at visual analogue scale
Serolology with immunoglobulins | 1 year before treatment, 4-6 weeks after treatment, 1 year after treatment
  Total and grass specific levels of IgE, IgG, IgG4, IgA in serum

CONTACTS AND LOCATIONS:
Overall Officials: Lars O Cardell, Professor, Principal Investigator — Karolinska Institutet
Locations (3):
- Sweden (3):
  - Skåne University Hospital, ENT department, Lund
  - Örebro University Hospital, Örebro
  - Karolinska University Hospital, ENT-department, Stockholm

IPD SHARING:
Plan to Share IPD: No